CLINICAL TRIAL: NCT05354492
Title: Evaluation of a New Program to Support Well-Being After Adversity
Brief Title: Evaluating a New Program for Successfully Coping With Adversity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wake Forest University (Other)
Collaborators: John Templeton Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00024316
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Trauma; Distress, Emotional; Psychological Distress
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Program Participant (Experimental): You will actively take part in the group program via Zoom with our program facilitators.
  Interventions: Other: Program to Support Well-Being after Adversity
- Program Wait List (No Intervention): You will be placed on a wait list to take part in the program.

INTERVENTIONS:
Other: Program to Support Well-Being after Adversity — You will be asked to meet on Zoom weekly for 6 weeks with our trained program facilitators along with the other 6-10 members of the intervention group. Meetings will last approximately 75-90 minutes each, and will involve a variety of discussions and activities related to navigating the changes you may face after experiencing a difficult life event. These sessions will be audio-recorded for research purposes and to ensure that facilitators are doing a good job delivering the program.
  Arms: Active Program Participant

SUMMARY:
You are invited to participate in a research study involving a new program designed to support people with navigating the changes that can happen after difficult life events. The program activities are aimed at helping you move forward and raise your well-being after experiencing one of life's challenges. This study should not be considered an alternative to any treatment or medication for any disorder or problem.

DETAILED DESCRIPTION:
Adversity is an inevitable part of human life and can potentially lead to great suffering. However, facing life's challenges also presents the opportunity for lasting and meaningful change. This phenomenon is referred to as posttraumatic growth (PTG) and has been defined as "positive psychological change experienced as the result of the struggle with highly challenging life circumstances" (Tedeschi & Calhoun, 2004). There are several existing psychosocial interventions (e.g., expressive writing) that have been shown to promote PTG, despite not being intentionally designed to do so. Additionally, there have been several interventions developed more recently that specifically target the cultivation of PTG, although many of them have not been extensively tested (Dolbier, Jaggars, & Steinhardt, 2010; Shakespeare-Finch et al., 2014). SecondStory 2.0 is an online group-format intervention that was augmented from the original program (SecondStory) which was designed to promote PTG and well-being in the face of adversity. SecondStory 2.0 incorporates narratives of moral exemplars who have overcome adversity, drawing from recent philosophical explorations that have highlighted the pedagogical functions of such exemplars (e.g. Zagzebski, 2017). This research has focused on their potential to model virtues that consistently characterize individuals who have overcome adversity (e.g. strength, vulnerability, wisdom, love, trust) (Brady, 2018). By including experiences of adversity in these exemplarist narratives, we can theoretically increase an individual's admiration for the exemplar, and in turn enable effective emulation while also broadening his/her understanding of the moral foundations of the human condition (Kidd, 2018).

This study will take place remotely via phone and zoom. The initial interview/screening will take place via an online Qualtrics survey (follow-up by phone with the study coordinator), and the intervention sessions will be held online via Zoom with our trained intervention facilitators (licensed therapists). We will also be providing intervention support via a text messaging platform called Mobile Coach. The messages will be the same for all of the participants, and they will all receive them at the same time point in the program. All of the questionnaires will be completed online via a link that will be texted and/or emailed to the participant. Once participants see an advertisement and reach out to our study coordinator about their interest in the study, they will be directed to complete an online prescreening survey via Qualtrics to assess their eligibility for study participation. The study coordinator will then review the online survey and complete the cognitive screener and mental health questions by phone. If participants are eligible after the phone screen with the study coordinator, they will be scheduled to do a safety assessment via phone with one of our study clinicians. Once participants are deemed eligible, they will complete the consent form and be randomized into one of two conditions: active program or control. If a participant is randomized into the control condition, they will be placed on a "wait list" to receive the intervention at a later date. If a participant is randomized into the active program condition, they will be given the schedule for the group sessions, and sent a Zoom link for participation. The group intervention sessions will be guided by our trained facilitators for 75-90 minutes weekly for six weeks. After week 6, participants who were in the active program group will be asked complete a feedback form, as well as to take part in a semi-structured group interview to determine the acceptability and feasibility of the program. They will then enter the follow-up period of the study. Regardless of condition, participants will complete a set of questionnaires at Weeks 0, 3, 6, 9, and 12.

After week 12, participants who were randomized to the control condition will receive access to a recorded version of the intervention online. The recorded version will include the intervention developer talking through the intervention content and materials on video. No study participants will be included in this video.

This data will help to inform us whether the new improvements made to the SecondStory protocol are effective in improving participants' overall well-being and response to trauma, and will guide any future changes made to the intervention protocol.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Have experienced trauma within the last 3 months to 5 years
* Feeling some level of subjective distress as a result of the trauma
* Read and understand English
* Have consistent access to the internet

Exclusion Criteria:

* Suicide risk
* Cognitive Impairment
* Diagnosed with a Psychotic Disorder
* Diagnosed with moderate to severe PTSD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Post-Traumatic Growth | 12 weeks
  We will use the Current-Standing Post-Traumatic Growth Inventory (C-PTGI)
Depression | 12 weeks
  We will use the Patient Health Questionnaire-8 (PHC-8)
Anxiety | 12 weeks
  We will use the Generalized Anxiety Disorder 7-item Scale (GAD-7)
Wellbeing | 12 weeks
  We will use Mental Health Checklist-Short Form (MHC-SF)
Vulnerability | 12 weeks
  We will use the Multidimensional Scale of Perceived Social Support (MSPSS)
Wisdom | 12 weeks
  We will use the Claremont Purpose Scale
Strength | 12 weeks
  We will use the State Hope Scale
Morality | 12 weeks
  We will use the Compassion Scale
Narrative Identity | 12 weeks
  We will code short qualitative responses for Personal Growth, Meaning-Making, Resolution, and Emotional Processing (Positive Reframing)

CONTACTS AND LOCATIONS:
Overall Officials: Eranda Jayawickreme, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States